CLINICAL TRIAL: NCT01730664
Title: Pharmacokinetics and Pharmacodynamics of Ertapenem in Patients With Tuberculosis
Brief Title: PK/PD of Ertapenem In Patients With TB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Jan-Willem C Alffenaar, PhD PharmD Clinical Pharmacologist, University Medical Center Groningen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ETB/V0.2
Record Dates: First submitted 2012-11-09; First posted 2012-11-21 (Estimated); Last update posted 2017-08-25 (Actual); Status verified 2017-08

CONDITIONS: PK of Ertapenem in TB Patients
Keywords: ertapenem; tuberculosis; pharmacokinetics
MeSH Terms: conditions — Tuberculosis | interventions — Ertapenem

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ertapenem (Experimental): single dose ertapenem
  Interventions: Drug: ertapenem

INTERVENTIONS:
Drug: ertapenem — single dose of 2000mg ertapenem IV

SUMMARY:
Rationale:

Treatment of multidrug or extensively drug resistant tuberculosis (MDR/XDR-TB) is a real challenge as failure in response to treatment and serious side-effects are frequently encountered. New, more effective drugs with less side effects are therefore urgently needed to solve this problem. Although several new drugs against TB are in the pipeline, physicians currently have limited treatment options for treatment of complicated MDR/XDR-TB cases. Therefore, drugs developed and labeled for other infectious diseases are evaluated for TB.

Objective:

The main objective of this prospective clinical trial is to evaluate pharmacokinetics of a standard dose (2000mg) of ertapenem in TB patients. This clinical trial will provide important information on PK of ertapenem in TB patients for future studies. Data can be used for limited sampling strategies for ertapenem based on a pharmacokinetic population model constructed from the full PK curves of the patients.

Study design:

A prospective pharmacokinetic study.

Study population: 12 TB patients.

Intervention: Single dose of 2000mg in a 30 minutes intravenous infusion.

Main study parameters/endpoints:

The pharmacokinetic parameters (Vd, Cl, AUC, etc) of ertapenem are the primary endpoints of the study. The T>MIC and AUC0-24h/Minimal inhibitory concentration (MIC) ratio are most likely the best predictive parameters for efficacy of ertapenem treatment and will be calculated for a range of M tuberculosis isolates.

ELIGIBILITY:
Inclusion Criteria:

* Patients with TB, with Mycobacterium tuberculosis (or M. africanum) by culture and / or molecular test
* Adults: from 18 years until 64 years of age

Exclusion Criteria:

-Contra-indications for ertapenem:

* There are few adverse effects of ertapenem. The only absolute contra- indication is a previous anaphylactic reaction to ertapenem or other β-lactam antibiotic.
* Renal Insufficiency, defined by a eGFR of 30ml/min
* Pregnancy
* HIV
* Body weight < 40 kg

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2017-01-26 (Actual); Primary Completion 2017-07-13 (Actual); Study Completion 2017-07-13 (Actual)

PRIMARY OUTCOMES:
AUC | first day
  main objective of this prospective clinical trial is to evaluate AUC of a standard dose (1000mg) of ertapenem in TB patients

SECONDARY OUTCOMES:
Safety: number of patients with organ dysfunction | day 1 and day 3
  renal function(eGFR) and liver enzymes(ALAT; ASAT)

OTHER OUTCOMES:
limited sampling strategies | day 1
  limited sampling strategies for ertapenem based on a pharmacokinetic population model constructed from the full PK curves of the patients.

CONTACTS AND LOCATIONS:
Locations (1):
- UMCG - Tuberculosis Center, Groningen, Netherlands

REFERENCES:
- [Background] Tremblay LW, Fan F, Blanchard JS. Biochemical and structural characterization of Mycobacterium tuberculosis beta-lactamase with the carbapenems ertapenem and doripenem. Biochemistry. 2010 May 4;49(17):3766-73. doi: 10.1021/bi100232q. PMID 20353175